CLINICAL TRIAL: NCT00656734
Title: A Phase 1, Open-Label, Multicenter Dose-escalation, Multidose Study of MDX1411 Administered Every 14 Days in Subjects With Advanced or Recurrent Clear Cell Renal Cell Carcinoma
Brief Title: Study of MDX-1411 Given Every 14 Days With Pre-medications to Subjects With Clear Cell Kidney Cancer.
Acronym: MDX1411-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1411-01; CA214-001 (Other: BMS)
Record Dates: First submitted 2008-04-03; First posted 2008-04-11 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Cancer
Keywords: Medarex Inc.
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDX 1411 (Experimental): Dose Escalation Cohorts
  Interventions: Biological: MDX 1411

INTERVENTIONS:
Biological: MDX 1411 — MDX-1411 (fully human monoclonal antibody) administered as an i.v. infusion for up to 5 doses per cycle, with a maximum of 17 cycles total

SUMMARY:
To determine the highest and safest tolerated dose of MDX-1411 for the treatment of clear cell renal cell carcinoma (Kidney cancer).

DETAILED DESCRIPTION:
Subjects will be assigned one dose upon enrollment and will continue with the same dose throughout the study. The maximum duration for the study is two and a half years for a total of 17 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of RCC with clear cell component
* Measurable disease
* Treated with up to 6 prior systemic therapies for advanced/recurrent disease or have become intolerant to a systemic therapy
* Subjects with treated brain metastases must be without magnetic resonance imaging (MRI) evidence of progression for at least 8 weeks and off steroids for at least 4 weeks to be eligible
* At least 28 days since the last chemotherapy
* At least 28 days before the first dose of MDX 1411 since any major surgery
* ECOG performance status 0-2
* No known positivity for human immunodeficiency virus (HIV), Hep B or C

Exclusion Criteria:

* Previous treatment with any other anti-CD70 antibody
* Active infection requiring i.v systemic therapy within 28 days before first dose
* Evidence of bleeding diathesis or coagulopathy
* Active autoimmune disease requiring immunosuppressive therapy
* Known current drug or alcohol abuse
* Any underlying medical condition which will make the administration of MDX 1411 hazardous
* Psychiatric illness or social situation that would preclude study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety profile of MDX 1411 | duration of study
Determine the maximum tolerated dose of MDX 1411 | duration of study

SECONDARY OUTCOMES:
Determine the best overall response rate (BORR) | Day 38-42 of each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon